CLINICAL TRIAL: NCT04256733
Title: A Pilot Study of Cough Reflex Desensitization for the Treatment of Cough Hypersensitivity Syndrome
Brief Title: Cough Desensitization Therapy for Cough Hypersensitivity Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Montana (Other)
Responsible Party: Principal Investigator, Laurie Slovarp, Associate Professor, University of Montana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 188-88
Record Dates: First submitted 2019-09-24; First posted 2020-02-05 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-08

CONDITIONS: Cough
Keywords: chronic cough; refractory chronic cough; cough hypersensitivity syndrome
MeSH Terms: conditions — Cough; Chronic Cough; cough hypersensitivity syndrome

STUDY DESIGN:
Intervention Model Description: One group will receive the placebo treatment while the second group receives the active treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blinded to group assignment (active treatment vs placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Supra-threshold capsaicin (Experimental): Participants will be exposed to progressively increasing concentrations of aerosolized capsaicin (the ingredient in chili peppers that makes them spicy, and a known cough stimulant) to stimulate an urge-to-cough. Participants will be coached to implement cough suppression strategies following each exposure.
  Interventions: Biological: Supra-threshold and progressive doses of diluted capsaicin via a Koko Digidoser nebulizer
- Sub-threshold capsaicin (Placebo Comparator): Participants will be exposed repeatedly to a single sub-threshold dose of aerosolized capsaicin through a nebulizer during treatment. This sub-threshold dose will elicit minimal or no urge-to-cough.
  Interventions: Biological: Sub-threshold doses of diluted capsiacin via a KoKo Digidoser nebulizer

INTERVENTIONS:
Biological: Supra-threshold and progressive doses of diluted capsaicin via a Koko Digidoser nebulizer — Participants will be exposured to increasing doses of aerosolized capsaicin (a known cough stimulant) through the Koko Digidoser nebulizer, while implementing behavioral cough suppression strategies. The concentration of capsaicin will increase incrementally as tolerated, as long as participants are still able to suppress cough. The concentration will never exceed 1000 micromolar. Participants will attend 6 treatment sessions and be given up to 12 exposures per treatment session. Participants will be encouraged to use cough suppression strategies outside of treatment sessions as much as possible to attempt to suppress cough.
  Arms: Supra-threshold capsaicin
Biological: Sub-threshold doses of diluted capsiacin via a KoKo Digidoser nebulizer — Participants will be repeatedly exposed to a sub-threshold dose of aerosolized capsaicin through the KoKo Digidoser nebulizer during treatment sessions. Participants will attend 6 treatment sessions and be given up to 12 exposures per treatment session. Participants will be encouraged to use cough suppression strategies outside of treatment sessions as much as possible to attempt to suppress cough.
  Arms: Sub-threshold capsaicin

SUMMARY:
The purpose of this study is to investigate a modified behavioral treatment for chronic cough due to cough hypersensitivity syndrome (CHS). This type of CC is a non-productive cough that is due, in part, to over-expression of transient receptor potential vanilliod (TRPV) receptors in the airway epithelium, which contribute to a dry cough elicited by typically non-tussive stimuli (e.g., cold air, smells) or by low doses of tussive stimuli (e.g., smoke). Currently available treatment options are limited to neuromodulator medications (e.g., gabapentin, amytriptiline) and behavioral cough suppression therapy (BCST), neither of which is 100% effective. The primary component of BCST is teaching patients to suppress their cough in the presence of an urge-to-cough. Studies have confirmed a reduction in cough sensitivity (as tested with inhaled capsaicin) following 1-4 weeks of successful cough suppression. However, patients with severe CHS are not able to suppress their cough in the presence of uncontrollable environmental stimuli and, hence, do not respond well to the therapy. The purpose of this study is to determine the potential of treating CHS by implementing BCST while stimulating cough with progressive concentrations of inhaled diluted aerosolized capsaicin. The investigators hypothesize this treatment will result in a reduction in cough-reflex sensitivity, cough-related quality of life, and cough frequency.

DETAILED DESCRIPTION:
The study will be a randomized, placebo-controlled, blinded study. It will take place in three phases, across 7 weeks.

WEEK 1: BASELINE TESTING AND TRAINING (approximate time = 1 hour).

1. Cough sensitivity testing: Standardized procedures that have been established and approved by the FDA will be used to determine cough sensitivity. Participants will inhale capsaicin vapor (a known cough stimulant) through a nebulizer with dosimeter, that delivers a specific dose of capsaicin in a mist form. They will inhale doubling doses of capsaicin mist from .49 micromolar to 1000 micromolar. The testing will be stopped when the investigators find the dose that causes five coughs or after giving the 1000 micromolar dose, whichever comes first. This testing will take approximately 30 minutes.
2. Urge-to-cough (UTC) testing: Participants be asked to report their UTC on a scale from 0 (no UTC) to 10 (maximum UTC) after each mist of capsaicin and after being presented with the following stimulants/tasks that cause some people to cough: perfume, bleach, vinegar, wood chips, laundry soap, cleaning wipe, deep and fast breath through the mouth, sustained voicing, reading a 55 word passage, and yelling a short phrase). This testing will take about 10 minutes.
3. Cough-related quality of life: Participants will complete the Leicester Cough Questionnaire which is a 23-item validated questionnaire designed to measure cough-related quality of life. It will take about 5 minutes.
4. Cough suppression training. Participants will be trained in cough suppression strategies. These strategies include 1) relaxed throat breathing where they inhale quickly through the nose and exhale through tightly pursed lips, and 2) cough suppression swallow, which involves swallowing saliva or a sip of water with as much effort as possible and while pressing hands together tightly. This training will take approximately 15 minutes.
5. Cough frequency testing: Participants will carry a small audio recording device with a small microphone that attaches to the participant's shirt for 24 hours. The recording device will be in a small carrying case (about half the size of a typical cell phone) that can clip to a belt or waistband. Participants will return the recording device to the investigators at or before the first treatment visit (see below). The audio recording will be analyzed by computer software that counts the number of coughs in the 24-hour period. (NOTE: The audio recording will not be listened to by any PERSON and the recording will be deleted after it is analyzed by the computer software.)

(Following baseline testing, participants will be randomly assigned to either the treatment group or placebo group.)

WEEKS 2-4: TREATMENT. Participants will attend treatment sessions twice per week for three weeks. Participants will use the breathing strategies following inhalation of either progressive doses of diluted capsaicin (experimental condition) or repeated exposures to a single sub-threshold concentration of diluted capsaicin (placebo condition). Participants will do this no more than twelve times per session. Each session will take approximately 45 minutes. If a participant misses a treatment session, the investigators will attempt to re-schedule that session. Each participant must complete at least five of treatment sessions to remain in the study.

WEEKS 5 AND 7: POST-TREATMENT TESTING. Outcome measures, as in the baseline phase, will be take at one-week and three-weeks post-treatment. The LCQ will be measured again at three-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Currently suffering from a cough that started at least 8 weeks ago
3. Have seen at least one physician for the cough and have received medical treatment without success
4. Normal chest x-ray, pulmonary function testing, and laryngoscopy (laryngoscopy completed by your physician or the speech-language pathologist)
5. Have undergone behavioral cough suppression therapy without full resolution of cough
6. Willing to take a pregnancy test before enrollment (if applicable)
7. Willing to use contraception during the study (if applicable)
8. Willing to sign an informed consent form

Exclusion Criteria:

1. Under 18 years of age
2. Currently a smoker of any substance
3. Pregnant or attempting to become pregnant
4. Diagnosed with a respiratory or pulmonary condition (e.g., asthma, COPD, emphysema, lung cancer, bronchitis)
5. Taken any of the following medications within the past month: lisinopril/Prinivil/Zestril, captopril/Capoten, enalapril/Epaned/Asotec, ramipril/Altace, benazepril/Lotensin, fosinopril/Monopril, moexipril/Univasc, perindopril/Aceonm, quinapril/Accupril, trandolapril/Mavik

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie J Slovarp, PhD, Principal Investigator — University of Montana
Locations (1):
- University of Montana, Missoula, Montana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Slovarp L, Reynolds JE, Bozarth-Dailey E, Popp S, Campbell S, Morkrid P. Cough desensitization treatment: A randomized, sham-controlled pilot trial for patients with refractory chronic cough. Respir Med. 2022 Mar;193:106739. doi: 10.1016/j.rmed.2022.106739. Epub 2022 Jan 15. PMID 35091204

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supra-threshold Capsaicin | Sub-threshold Capsaicin
Started | 11 | 8
Completed | 8 | 6
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supra-threshold Capsaicin | Sub-threshold Capsaicin | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.25 (15.9) | 66 (13.6) | 63.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 8 | 19
Leicester Cough Questionnaire (LCQ) [Mean (Standard Deviation); unit: units on a scale] — The LCQ is a 19-item patient-report questionnaire that measures the impact of cough on quality of life. The questions are divided into Psychological, Physical, and Social subscales which are an average of the questions that make up each subscale. The range for each subscale is 1-7. The subscale scores are summed to get a total LCQ score, which can range from 3-21. A higher score indicates less impact on quality of life.
  units on a scale | 12.65 (3.11) | 12.43 (2.69) | 12.56 (2.83)
Urge-to-cough (UTC) test: UTC sum [Mean (Standard Deviation); unit: units on a scale] — During UTC testing, participants are exposed to various scents and various vocal and breathing tasks (12 tasks in total). After each task, they report the maximum UTC they felt during the task on a scale from 0 (no UTC) to 10 (maximum UTC). The UTC scores for each task are summed for a single score. This results in a possible UTC score of 0 (no UTC on any tasks) to 120 (maximum UTC on every task).
  units on a scale | 18.19 (15.67) | 14.67 (11.50) | 16.68 (13.65)
Urge-to-cough (UTC) test: cough frequency sum [Mean (Standard Deviation); unit: sum cough frequency] — During UTC testing, participants are exposed to various scents and complete various vocal and breathing tasks. They are instructed to let their body react naturally after each task and to NOT try to suppress their cough. The number of coughs elicited during each task is recorded. The final score is a sum of the cough frequency for each task.
  sum cough frequency | 14.38 (20.12) | 9.67 (11.76) | 12.36 (16.64)

OUTCOME MEASURES:

1. Primary Outcome: Leicester Cough Questionnaire (LCQ)
Description: The Leicester Cough Questionnaire (LCQ) is a 19-item validated patient-report questionnaire that measures the impact of cough on quality of life. It takes about 5 minutes to complete and results in three domain scores (Social, Psychological, and Physical), and one Total score. Domain scores are averages of the questions that make up each domain. Minimum and maximum domain scores are 1 and 7, respectively. The domain scores are summed to determine the Total score, which can range from 3 to 21. A higher score means less impact on quality of life. The change in LCQ was determined by subtracting the Total LCQ score at baseline from the Total LCQ score at 3 weeks post-treatment. A positive LCQ change score indicates an improvement.
Time Frame: The LCQ will be measured before treatment and three weeks following treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supra-threshold Capsaicin | Sub-threshold Capsaicin
Number analyzed (Participants) | 8 | 6
score on a scale | 3.2 (1.78) | 2.06 (2.48)
Statistical Analysis 1: Comparison: Supra-threshold Capsaicin vs Sub-threshold Capsaicin; Test type: Superiority; p = .23, Mixed Models Analysis

2. Secondary Outcome: Urge-to-Cough Testing
Description: Urge-to-cough (UTC) testing involves presenting participants to various scents and vocal and breathing tasks (12 tasks in total) and asking them to rate their maximum perceived UTC on a scale from 0 (no UTC) to 10 (maximum UTC). The UTC score for each testing session is the sum of the the UTC scores from each individual task. This results in a possible score range from 0 (no UTC on any tasks) to 120 (score of 10 on every UTC task). UTC change is determined by subtracting the UTC score on each task at baseline from the UTC score for each task at 3 weeks post-treatment and then summing those scores. A negative UTC change score indicates the UTC score was lower post-treatment relative to baseline, which indicates an improvement.
Time Frame: Urge-to-cough will be measured before treatment and three weeks following the final treatment session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supra-threshold Capsaicin | Sub-threshold Capsaicin
Number analyzed (Participants) | 8 | 6
units on a scale | -13.75 (10.45) | -8.8 (10.34)
Statistical Analysis 1: Comparison: Supra-threshold Capsaicin vs Sub-threshold Capsaicin; Test type: Superiority; p = .57, Mixed Models Analysis

3. Secondary Outcome: Urge-to-Cough Testing: Cough Frequency
Description: During UTC testing, participants are exposed to various scents and vocal and breathing tasks and the number of coughs elicited during and immediately following each task are counted. A cough frequency score for each testing session is the sum of the number of coughs counted during each task. Change in cough frequency is calculated by subtracting the baseline cough frequency from the 3 week post-treatment cough frequency. A negative score indicates cough frequency was less after treatment, which indicates an improvement.
Time Frame: Baseline and 3 weeks post-treatment
Measure: Mean (Standard Deviation); unit: coughs
Arm/Group | Supra-threshold Capsaicin | Sub-threshold Capsaicin
Number analyzed (Participants) | 8 | 6
coughs | -14.00 (20.10) | -6.33 (9.16)
Statistical Analysis 1: Comparison: Supra-threshold Capsaicin vs Sub-threshold Capsaicin; Test type: Superiority; p < .0001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the treatment period and for three weeks following the treatment period for a total of 9 weeks.
Arm/Group | Supra-threshold Capsaicin | Sub-threshold Capsaicin
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 0/11 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT04256733/Prot_SAP_000.pdf